CLINICAL TRIAL: NCT03380260
Title: Investigating Neural Processing of Social Stimuli: Investigating a Neurobehavioral Mechanism of Paranoia
Brief Title: Investigating Neural Processing of Social Stimuli
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas at Dallas (Other)
Responsible Party: Principal Investigator, Amy Pinkham, Associate Professor, The University of Texas at Dallas
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: 17-44
Record Dates: First submitted 2017-12-11; First posted 2017-12-21 (Actual); Last update posted 2021-04-28 (Actual); Status verified 2021-04

CONDITIONS: Healthy Adults

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Paranoia Induction (Experimental): Behavioral procedure involving social exclusion and negative feedback to induce paranoia
  Interventions: Behavioral: Paranoia Induction
- Control Condition (No Intervention): No manipulation of paranoid ideation

INTERVENTIONS:
Behavioral: Paranoia Induction — Behavioral procedure involving social exclusion and negative feedback to induce paranoia
  Arms: Paranoia Induction

SUMMARY:
The primary goal of the present study is to test whether neural activity in brain regions associated with processing threat and social stimuli may underlie paranoid thinking.

DETAILED DESCRIPTION:
Paranoia is a prominent symptom of psychosis that occurs in several other diagnoses, as well as the general population, and that is associated with significant distress and impairment. Previous research suggests that increased baseline activity of the amygdala and related neural circuits may serve as a mechanism for paranoid ideation. This exploratory study will use a paranoia induction procedure in healthy individuals who vary in pre-existing levels of paranoid ideation to test whether increases in self-reported paranoia are accompanied by increases in resting cerebral blood flow (CBF), decreased stimulus-driven neural activity in social processing networks, and increased behavioral perceptions of untrustworthiness.

Participants will be randomly assigned to participate in a paranoia induction procedure or a control condition and will then complete neuroimaging and behavioral assessments.

ELIGIBILITY:
Inclusion Criteria:

* between the ages of 18 and 55

Exclusion Criteria:

* current psychiatric diagnosis
* current use of psychotropic medications
* history of head trauma with loss of consciousness for more than 15 minutes
* presence of neurological or neurodegenerative disorder
* sensory impairments that preclude assessment
* presence of intellectual disability
* contraindications for MRI (e.g., metallic implants or pregnancy)

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 70 (Actual)
Dates: Start 2017-06-01 (Actual); Primary Completion 2019-04-01 (Actual); Study Completion 2019-04-01 (Actual)

PRIMARY OUTCOMES:
Resting cerebral blood flow (CBF) | CBF measurements will be obtained during the study visit and will last approximately 9 minutes.
  CBF in amygdala and related neural circuits

SECONDARY OUTCOMES:
Amount of Neural Activity | Measurements will be obtained during the study visit and will last approximately 25 minutes.
  Task-related activation of amygdala and related neural circuits measured with blood-oxygenation-level-dependent imaging
Ratings of Trustworthiness | Data will be obtained during the study visit and will last approximately 12 minutes.
  Behavioral perceptions of the trustworthiness of others
Self-reported paranoid ideation | Data will be obtained during the study visit and will last approximately 5 minutes.

CONTACTS AND LOCATIONS:
Overall Officials: Amy Pinkham, PhD, Principal Investigator — The University of Texas at Dallas
Locations (1):
- Advanced Research Imaging Center, The University of Texas Southwestern Medical School, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No